CLINICAL TRIAL: NCT05545384
Title: Immediate Versus Delayed Treatment With Azathioprine or Rituximab in Anti-myelin Oligodendrocytes Glycoprotein (Anti-MOG) Antibodies Associated Acute Demyelinating Syndromes in Children: a Randomized Controlled Clinical Trial
Brief Title: Immediate Versus Delayed Treatment With Azathioprine or Rituximab in Anti-MOG Antibodies Associated Acute Demyelinating Syndromes in Children: a Randomized Controlled Clinical Trial
Acronym: IDAR
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP211057; 2022-002385-32 (EudraCT Number)
Record Dates: First submitted 2022-09-06; First posted 2022-09-19 (Actual); Last update posted 2025-04-07 (Actual); Status verified 2025-03

CONDITIONS: Acute Demyelinating Syndrome
Keywords: acute demyelinating syndrome
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: This is a multicentre, randomized controlled, open-labelled, parallel group study.
Masking Description: The adjudication committee is responsible the evaluation of all relapses reported during the the follow-up period. Relapses assessments will use blinded data and will be performed in real time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Immediate Azathioprine (1st attack) (Experimental): Treatment will be started at 2mg/kg or at 1mg/kg if the patient has a partial activity which would be increased slowly according the 6-TGN activity and clinical and biological tolerance at Week 2 for patient with partial activity or M1 for patient without TPMT activity deficit.
  Only for patient with partial deficit and whose 6-TGN activity is low, azathioprine would be increased at 3mg/kg/d at Week 6 and without exceeding a total daily dose of 150 mg.
  Interventions: Drug: Immediate Azathioprine (1st attack)
- Immediate Rituximab (1st attack) (Experimental): Once the inclusion criteria are validated, the first injection will be performed according to the injection protocol (Annex 4). Fifteen day later, the second injection will be performed.
  The next visit during a consultation with PI or his collaborators will be scheduled 1 week ± 2 days later, and patients will be advised to contact the PI if any neurologic symptoms or symptoms of adverse event occurs in the meantime.
  Interventions: Drug: Immediate Rituximab (1st attack)
- Standard Care: delayed treatment (2nd attack) (Active Comparator): Patients will be treated according to standard of care after their 1st attack. In case of relapse:
  * before 3 months, IV methylprednisolone (30 mg/kg/j not exceeding 1g/day) will be administered for 3 days. There won't be any change of the initial treatment which will be pursued.
  * after 3 months, IV methylprednisolone (30 mg/kg/j not exceeding 1g/day) will be administered for 3 days with an oral relay of prednisolone (1mg/kg/day not exceeding 60 mg/day) during 3 months with then a slowly tapered dose (reduction of 25% every week for 4 weeks). Azathioprine or Rituximab might be proposed as per local clinician experience
  Interventions: Drug: Standard of care

INTERVENTIONS:
Drug: Immediate Azathioprine (1st attack) — Patients randomized in Immediate Azathioprine group will benefit from immediate treatment with azathioprine. Treatment will be started at 2mg/kg or at 1mg/kg if the patient has a partial activity which would be increased slowly according the 6-TGN activity and clinical and biological tolerance at Week 2 for patient with partial activity or M1 for patient without TPMT activity deficit.
  Only for patient with partial deficit and whose 6-TGN activity is low, azathioprine would be increased at 3mg/kg/d at Week 6 and without exceeding a total daily dose of 150 mg.
  Arms: Immediate Azathioprine (1st attack)
Drug: Immediate Rituximab (1st attack) — Patients randomized in Immediate Rituximab group will benefit from immediate treatment with rituximab. Rituximab 375mg/m2 IV will be given at D1 and D15 and repeat every 6 months for 2 years.
  Once the inclusion criteria are validated, the first injection will be performed according to the injection protocol (Annex 4). Fifteen day later, the second injection will be performed.
  The next visit during a consultation with PI or his collaborators will be scheduled 1 week ± 2 days later, and patients will be advised to contact the PI if any neurologic symptoms or symptoms of adverse event occurs in the meantime.
  Arms: Immediate Rituximab (1st attack)
Drug: Standard of care — Patients in this group will be treated according to standard care
  Arms: Standard Care: delayed treatment (2nd attack)

SUMMARY:
Among all non viral encephalitis, myelin oligodendrocytes glycoprotein antibody associated diseases (MOGAD) are the second most frequent diagnosis in children. Risk of relapses varies according to studied cohorts and cognitive and academic difficulties are more and more detected in children without knowing if these sequelae are related to the first attack or relapses. The hypothesis is that earlier treatment would induce reduction of sequelae after the first attack and the number of relapses which would be also associated with a subsequent reduction of disability occurrence on the long term.

DETAILED DESCRIPTION:
Acquired Demyelinating Syndrome (ADS) are rare immune-mediated central nervous system (CNS) disorders that contribute to significant neurological morbidity in Europe and worldwide. ADS can affect adult and children, and the clinical spectrum is heterogenous. It begins as monophasic diseases, as often observed in acute demyelinating encephalomyelitis (ADEM), optic neuritis (ON) and transverse myelitis (TM); or as multiphasic disease with relapses such as multiple sclerosis (MS) or neuromyelitis optica spectrum disorders (NMOSD).

MOG-Abs-ADS are a frequent disease in children with ADS with specific clinical and MRI pattern.

Recently, myelin oligodendrocyte glycoprotein (MOG) antibodies (MOG-Abs) have been found implicated in ADS affecting children with a frequency up to 30%-45% according to tested cohorts.

Studies have shown that in MOG-Abs positive ADS, the most frequent clinical phenotype in children are ADEM-like presentations (ADEM, ADEM-optic neuritis, multiphasic demyelinating encephalomyelitis (MDEM) and encephalitis) and optic neuritis (ON). These presentations may vary according to the age and young children < or = 10 years old, most often, present with ADEM, whereas optic neuritis is the most common feature in children older than 10 years of age. Fewer patients present with myelitis, brainstem features, or the more recently described encephalitis with steroid-responsive seizures11.

Cerebro-spinal fluid parameters are normal in most patients, although up to 50% had pleiocytosis or increased protein levels. Oligoclonal bands were present in only 10% of patients and their presence in the context of relapsing disease would rather suggest MS 5.

MRI lesions are particular in MOG-Abs positive ADS: lesions are distributed in the cortex, subcortical region, deep white matter, brainstem, thalamus, basal ganglia and are characterized by poor demarcation and large size. These features have been found particularly in ADEM and MDEM and when compared to MOG-Abs negative ADS, large, hazy and bilateral lesions, an absence of small lesions and/or well-defined lesions, and involvement of more anatomical areas, often with longitudinally extensive transverse myelitis have been described. Absence of corpus callosal lesions, presence of cerebellar peduncle and leukodystrophy-like lesions were also observed in MOG-Ab-positive cases. MOG-Ab-associated optic neuritis is characterized on MRI by optic nerve head swelling, retrobulbar involvement, a long lesion length and, frequently, bilateral involvement.

MOG-Abs-ADS are highly relapsing and may be associated with disabilities More than 40% of MOGAD relapse mimicking diseases such as MS or anti aquaporin 4 (AQP4-Abs) positive NMOSD with an higher relapse rate 6. In the French national retrospective study on anti-MOG-Abs positive ADS, it was observed that relapse occurred in 46% of included children with a median time of 10 months (range :1-305 months) after onset, results that are in line with studies in other European countries 9.

Relapses are frequently observed during steroid weaning or within 2 months of steroid withdrawal 7, 9, 16-18. Most relapses occur in adults who are being treated with prednisolone <10 mg daily (range 0-25 mg) or in children who are receiving prednisolone <0.5 mg/kg daily. The duration of treatment might also be important. Patients whose treatment lasts for less than 3 months are twice as likely to relapse as those who are treated for longer, suggesting the need for a biomarker for the response to treatment. Several studies suggest that relapses occur in patients who remain seropositive despite treatment particularly in patients who often have high initial antibody titres.

Studies in optic neuritis, the most common neurological symptom in MOG-Abs-ADS have demonstrated that severe damage to the optic nerve can be observed in MOG-Ab-associated disorders. The observed damage seems to be driven by the frequency of attacks in patients who recover from the initial episode suggesting the need of long term treatment. Moreover, although most patients with MOG-Ab-associated disease recover well from attacks, it has also been shown that up to 45% can be left with severe disability. Importantly, >70% of this disability results from the onset attack, suggesting that there is room for improvement in the acute management of MOG-Ab-associated disease, and that time to treatment might be important for the prevention of permanent disability.

Recently, Bicêtre's hospital medical team have performed a multi-national collaborative study on 102 children with relapsing MOG-Abs-ADS (RADS) through a European Consortium coordinated by the coordinator of this project. In that study, it was observed that although the majority of children had low level clinical disability, 20% of affected children had cognitive impairment and investigators confirmed these results in the national cohort study where they have observed that age at onset < or = 10 years (OR, 3.72, 95%CI 1.19-11.64; p=0.024), ADEM at onset (OR 52.5, 95%CI 5.97-461.4; p<0.001), and deep grey matter lesions (OR, 17.33 95%CI 3.87-77.72; p<0.001) were associated to the presence of cognitive difficulties.

Studies on prospective treatment of MOGAD are rare and current treatment is based on clinical experience with similar antibody-mediated diseases, such as AQP4-Abs positive NMOSD. Corticosteroids, intravenous immunoglobulin, immunosuppressive drugs (such as mycophenolate mofetil, azathioprine and methotrexate) and rituximab are actually used and are associated with a reduction in annual relapse rate. By contrast, immunomodulatory treatments for MS, such as interferon-β and glatiramer acetate, are ineffective. In a study of children and adults in Australia, maintenance treatment with oral prednisolone was associated with fewer treatment failures than were other treatment modalities, whereas in the European collaborative retrospective study of children with MOG-Abs, investigators were able to confirm that all treatment modalities reduced annualized relapse rates but had limited effects on disability. Due to the immense vacuum in the treatment strategies, investigators have also established established an European consensus on treatment and emphasized on the absolute need for a randomized controlled treatment trials to find an optimal therapeutical strategy in order to reduce risk of sequelae after the first attack and relapses that could reduce disabilities.

ELIGIBILITY:
Inclusion Criteria:

* Children < 18 years old and ≥ 6 years old at baseline
* Children weight ≥ 20 kg
* All ADS with confirmed anti-MOG-Abs at onset including any acute neurologic symptom with a duration of more than 24H of inflammatory causes (including optic neuritis, transverse myelitis, rhombencephalitis, ADEM, NMOSD) Without any previous treatment other than steroids
* Informed consent signed by both parents and the child
* Expanded Disability Status Scale (EDSS) < 5.5
* Affiliated to French social security regime

Exclusion Criteria:

* Current infection with SARS-COV2 (positive PCR)
* Any prior allergy to azathioprine or rituximab with hypersensitivity to active substances, murine proteins or to any of the excipients.
* Any prior history of uncontrolled cancer during the last 2 years
* Uncontrolled infections (Hepatitis B, C and HIV)
* Any prior history of cardiac dysfunction and/or hypertension
* Any progressive or non-relapsing form demyelinating diseases
* Any previous treatment with natalizumab, daclizumab, fingolimod, methotrexate, cyclosporine, mycophenolate mofetil, rituximab in the last 6 months, or determined by the treating physician to have residual immune suppression from these or other immunosuppressive treatments
* CD4+, CD8+, or CD19+ absolute cell count, wbc, neutrophiles in blood at screening below lower limits of normal (LLN)
* Creatinine>30µmol/L
* Platelets <70 000mm3
* Haemoglobin < 8g/dL
* Acute renal insufficiency (clearance < 30 ml/min)
* Prior documented history of hemostase perturbation (TP and/or TCA more than twice of the witnesse's TP and/or TCA)
* Prior documented history of increased liver enzyme level (ASAT and/or ALAT) > 2N.
* TP <70%
* Total bilirubin > 2N
* Any patient with allopurinol treatment and immunosupressive treatment with concomitant use of xanthine oxidase inhibitors (e.g. allopurinol, oxipurinol/thiopurinol, febuxostat)
* Patients with two inactive TPMT or NUDT15 alleles (homozygous deficient or double heterozygote)
* Pregnancy or lactating woman or wish for future pregnancy
* Refusal to have a highly effective contraception during traitment and for one year (12 months) after the end of the experimental treatment
* participation to another interventional study within 5 half-lives prior to baseline.
* Active, severe infections (including tuberculosis, HBV and HCV, HIV, herpes, VZV, EBV and CMV)
* Psychosis not controlled by treatment
* Patients with Lesch Nyhan syndrome
* Pheochromocytoma
* Scleroderma
* Untreated peptic ulcer
* Myasthenia gravis
* Any other medical illness or disability that, in the opinion of the investigator, would compromise effective trial participation

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
annualized relapse rate (ARR) at 24 months | at 24 months
  To compare the efficacy of immediate (at first attack) azathioprine (AZA) or rituximab (RTX) treatment in children with MOG antibodies positive diseases with delayed treatment (at second attack), on the annualized relapse rate at 24 months.

SECONDARY OUTCOMES:
Annualized relapse rate at 12 months | at 12 months
  Evaluate the efficacy of immediate treatment with delayed treatment
Time to first relapse (2nd attack) will be defined as time from randomization to the date of first relapse, with right-censoring in case of loss of follow-up | through study completion, an average of 2.5 years
  Evaluate the efficacy of immediate treatment with delayed treatment
Percentage of patients free of relapses over 24 months | through study completion, an average of 2.5 years
  Evaluate the efficacy of immediate treatment with delayed treatment
Motor disability outcome will be assessed with Expanded Disability Status Scale (EDSS) score | through study completion, an average of 2.5 years
  Evaluate the efficacy of immediate treatment with delayed treatment. The EDSS is an ordinal scale used for assessing neurologic impairment based on a neurological examination. It consists of scores in each of seven central functional systems (FSs) that are then combined to determine the EDSS steps (ranging from 0 (normal) to 10 (death due to MS)). The FSs are Visual, Brain Stem, Pyramidal, Cerebellar, Sensory, Bowel & Bladder, and Cerebral functions. EDSS is a widely used and accepted instrument to evaluate disability status at a given time and, longitudinally, to assess disability progression in clinical studies in MS other MOG-Abs-ADS related studies.
Visual Acuity, Optical Coherence Tomography | at 3, 6, 12 and 24 months
  Evaluate the efficacy of immediate treatment with delayed treatment.
Cognitive function: Wechsler Intelligence Scale for Children (WISC)-5 | at 6 and 24 months
  Evaluate the efficacy of immediate treatment with delayed treatment.
Fatigue Severity Scale (FSS) | at 6, 12, 18 and 24 months
  Evaluate the efficacy of immediate treatment with delayed treatment.
Cumulative number of new or newly enlarged lesions detected on T2-weighted MRI and of T1 gadolinium enhancing lesions | at 6, 12, 18 and 24 months
  Evaluate the efficacy on MRI outcomes

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU Besançon, Besançon
  - CHU Bordeaux, Bordeaux
  - CHU Brest, Brest
  - HCL de Bron, Bron
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHRU Lille, Lille
  - CHU Monptellier, Montpellier
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse Purpan, Toulouse